CLINICAL TRIAL: NCT02783807
Title: Clinical Equivalency Validation Protocol Eyenez v200 and Volk Pictor Ret1
Brief Title: Clinical Equivalency Validation Protocol Clinical Equivalency Eyenez Retina Camera v200 and Optomed Smartscope M5 EY3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eyenez LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 101
Record Dates: First submitted 2016-05-18; First posted 2016-05-26 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-05

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Eyenez Retinal Camera v200 (Experimental): Retinal images from Eyenez Retinal Camera v200 of healthy and diseased subjects
  Interventions: Device: Eyenez Retinal Camera v200
- Volk Pictor Ret 1 (Active Comparator): Retinal images from Volk Pictor Ret 1 of healthy and diseased subjects
  Interventions: Device: Volk Pictor Ret 1

INTERVENTIONS:
Device: Eyenez Retinal Camera v200
  Arms: Eyenez Retinal Camera v200
Device: Volk Pictor Ret 1
  Other Names: Optimed Smartscope M5 EY3
  Arms: Volk Pictor Ret 1

SUMMARY:
This prospective equivalency study compares the performance of two Ophthalmic Cameras, the Eyenez Retina Ophthalmic Camera v200 (OC) and the Optomed Smartscope M5 EY3 (OP). Trained technicians will take pictures of the same patients' retinas and the quality of the photos will be evaluated. The study includes healthy patients and patients with a spectrum of retinal diseases. The study requires that technicians take pictures of the retinas of adult patients between 18 and 80 years of age using both the OC and OP. The pictures will be reviewed and compared by a central reader/Ophthalmologist, who will determine if the OC is equivalent to the OP, based on the quality of the images

DETAILED DESCRIPTION:
Subjects (patients) will be recruited via word of mouth.

The study duration will be approximately 1-2 weeks, assuming a recruitment rate of 15 subjects per week. The images will be recorded within 15 minutes and will involve minimal disruption to the clinical workflow.

In the Study Environment setting (Foothill Medical Offices), the User Interface will be evaluated by comparing retinal pictures taken with subject device OC and predicate device OP.

Patient subjects will be given an Information and Consent Form to complete prior to the study

The technicians employed by Foothill Eye Clinic will operate the device on patient participants by taking a retinal picture using OC.

The technicians will use the predicate device OP to take retinal pictures.

The Ophthalmologist will compare the results with the pictures taken by OC and OP. The Ophthalmologist will be blinded to what picture was taken by which camera and record his assessment of the quality for each picture.

Patient subjects will receive a standard of care exam with or without dilation.

ELIGIBILITY:
Healthy subjects Inclusion Criteria:

* Written Informed Consent
* Male or female
* Age ≥ 18 years and ≤80 years
* Normal Retina

Healthy subjects Exclusion Criteria:

* Glaucoma
* Limited Ability for Agreement
* Spectrum of retinal diseases
* Subjects that may have been exposed to retinal photography in the past 24 hours prior to the study visit or plan to have retinal photography in the 24 hours after the study visit

Diseased subjects Inclusion Criteria:

* Written Informed Consent
* Male or female
* Age ≥ 18 years and ≤80 years
* Spectrum of retinal diseases

Diseased subjects Exclusion Criteria:

* Normal Retina
* Limited Ability for Agreement
* Subjects that may have been exposed to retinal photography in the past 24 hours prior to the study visit or plan to have retinal photography in the 24 hours after the study visit

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-10; Primary Completion 2016-03 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Clinical Evaluation of Retina Camera Images from both Healthy and Diseased Subjects | up to 1 week
  At least 90% of retinal camera images from both retinal cameras will be equivalent

CONTACTS AND LOCATIONS:
Overall Officials: Mark Kislinger, PhD MD, Principal Investigator — Eyenez LLC

IPD SHARING:
Plan to Share IPD: Yes
510k Submission